CLINICAL TRIAL: NCT02351427
Title: Bortezomib With Steroid Pulse Therapy for Acute Cellular Rejection in Kidney
Brief Title: Bortezomib With Steroid Pulse Therapy for Acute Cellular Rejection in Kidney Transplantation
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Su-Kil Park, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-1223
Record Dates: First submitted 2015-01-27; First posted 2015-01-30 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Kidney Transplantation
MeSH Terms: interventions — Bortezomib; Steroids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bortezomib (Active Comparator): Bortezomib (subcutaneous) 1.3mg/m2 on day 1, 4 and 7
  with
  Steroid - Methylprednisolone (intravenous) Day 1 - 7: 500 mg/500 mg/500 mg/250 mg/250 mg/125 mg/125 mg After day 7: prednisolone (oral) 30 - 60 mg, then taper the dosage
  Interventions: Drug: Bortezomib; Drug: Steroid
- Steroid (Active Comparator): Steroid - Methylprednisolone (intravenous) Day 1 - 7: 500 mg/500 mg/500 mg/250 mg/250 mg/125 mg/125 mg After day 7: prednisolone (oral) 30 - 60 mg, then taper the dosage
  Interventions: Drug: Steroid

INTERVENTIONS:
Drug: Bortezomib — In one group, investigators administer bortezomib and steroid to manage acute cellular rejection in kidney transplantation, and compare the results with another group in which only steroid was administered.
  Other Names: Velcade
  Arms: Bortezomib
Drug: Steroid — Investigators administer steroid in both groups for conventional treatment of acute cellular rejection.

SUMMARY:
The purpose of this study is to determine whether bortezomib is effective in the treatment of acute cellular rejection after kidney transplantation.

DETAILED DESCRIPTION:
When acute cellular rejection occurred in kidney allograft, investigators administer high dose steroid. However, there is insufficient effect in about 20-30%. Bortezomib acts not only on plasma cells, but also T cells, B cells and dendritic cells. In addition, bortezomib is relatively safe drug compared to thymoglobulin which investigators use in the cases of steroid failure. Therefore, investigators administer bortezomib with steroid in one group, and compared the group with the other group in which conventional steroid treatment is done.

ELIGIBILITY:
Inclusion Criteria:

* living donor kidney transplantation recipients
* patients who were performed kidney biopsies because of laboratory and clinically suspected rejection
* Biopsy proven acute cellular rejection (Banff I - IIA) with C4d negative
* Single luminex panel reactive antibody (PRA) I & II mean fluorescent intensity (MFI) < 3000

Exclusion Criteria:

* patients who received other major organ transplantation
* combined with urinary tract infection or obstruction
* combined with acute antibody mediated rejection
* poor compliance

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-02; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Serum creatinine | Day 14
  Investigators measure patients' serum creatinine at day 14.

SECONDARY OUTCOMES:
Incidence of steroid failure | Day 7
  Steroid failure is defined as serum creatinine at day 8 ≥ serum creatinine at day 0.
Serum creatinine | Month 1
  Investigators measure patients' serum creatinine at month 1.
Infection | Until 1 year after intervention
  Infection as measured by clinical, laboratory and microbiological data
Recurrence of Rejection | Until 1 year after intervention
  Recurrence of rejection as measured by clinical and laboratory data with graft biopsy.

CONTACTS AND LOCATIONS:
Overall Officials: Su-Kil Park, M.D., PhD, Principal Investigator — Division of Nephrology, Department of Internal Medicine, Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Background] Lemy A, Toungouz M, Abramowicz D. Bortezomib: a new player in pre- and post-transplant desensitization? Nephrol Dial Transplant. 2010 Nov;25(11):3480-9. doi: 10.1093/ndt/gfq502. Epub 2010 Sep 8. PMID 20826741
- [Background] Walsh RC, Alloway RR, Girnita AL, Woodle ES. Proteasome inhibitor-based therapy for antibody-mediated rejection. Kidney Int. 2012 Jun;81(11):1067-74. doi: 10.1038/ki.2011.502. Epub 2012 Feb 15. PMID 22336990
- [Background] Tzvetanov I, Spaggiari M, Joseph J, Jeon H, Thielke J, Oberholzer J, Benedetti E. The use of bortezomib as a rescue treatment for acute antibody-mediated rejection: report of three cases and review of literature. Transplant Proc. 2012 Dec;44(10):2971-5. doi: 10.1016/j.transproceed.2012.02.037. PMID 23195008
- [Background] Schmidt N, Alloway RR, Walsh RC, Sadaka B, Shields AR, Girnita AL, Hanseman DJ, Woodle ES. Prospective evaluation of the toxicity profile of proteasome inhibitor-based therapy in renal transplant candidates and recipients. Transplantation. 2012 Aug 27;94(4):352-61. doi: 10.1097/TP.0b013e318257acf6. PMID 22836132
- [Background] Hu X, Xu J, Sun A, Shen Y, He G, Guo F. Successful T-cell acute lymphoblastic leukemia treatment with proteasome inhibitor bortezomib based on evaluation of nuclear factor-kappaB activity. Leuk Lymphoma. 2011 Dec;52(12):2393-5. doi: 10.3109/10428194.2011.593271. Epub 2011 Jul 12. No abstract available. PMID 21745166
- [Background] Kim SJ, Yoon DH, Kang HJ, Kim JS, Park SK, Kim HJ, Lee J, Ryoo BY, Ko YH, Huh J, Yang WI, Kim HK, Min SK, Lee SS, Do IG, Suh C, Kim WS; Consortium for Improving Survival of Lymphoma (CISL) investigators. Bortezomib in combination with CHOP as first-line treatment for patients with stage III/IV peripheral T-cell lymphomas: a multicentre, single-arm, phase 2 trial. Eur J Cancer. 2012 Nov;48(17):3223-31. doi: 10.1016/j.ejca.2012.06.003. Epub 2012 Jul 4. PMID 22770877
- [Background] Zain JM, O'Connor O. Targeted treatment and new agents in peripheral T-cell lymphoma. Int J Hematol. 2010 Jul;92(1):33-44. doi: 10.1007/s12185-010-0614-9. Epub 2010 Jun 10. PMID 20535594
- [Background] Arnulf B, Pylypenko H, Grosicki S, Karamanesht I, Leleu X, van de Velde H, Feng H, Cakana A, Deraedt W, Moreau P. Updated survival analysis of a randomized phase III study of subcutaneous versus intravenous bortezomib in patients with relapsed multiple myeloma. Haematologica. 2012 Dec;97(12):1925-8. doi: 10.3324/haematol.2012.067793. Epub 2012 Jun 11. PMID 22689676
- [Result] Everly MJ, Everly JJ, Susskind B, Brailey P, Arend LJ, Alloway RR, Roy-Chaudhury P, Govil A, Mogilishetty G, Rike AH, Cardi M, Wadih G, Tevar A, Woodle ES. Bortezomib provides effective therapy for antibody- and cell-mediated acute rejection. Transplantation. 2008 Dec 27;86(12):1754-61. doi: 10.1097/TP.0b013e318190af83. PMID 19104417